CLINICAL TRIAL: NCT01819688
Title: Surgical Stress Induced Insulin Resistance and Cytokine Response After Laparoscopic Compared to Open Liver Resection
Brief Title: Surgical Stress After Laparoscopic Compared to Open Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Chun-Yan Yan, M.D. , Ph.D, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20120704; (1)2009R50040 (2)LY12H02005 (Other Grant/Funding Number: (1) Foundation of Science and Technology Department of Zhejiang (2)Zhejiang Provincial Natural Science Foundation)
Record Dates: First submitted 2013-03-20; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Insulin Resistance
Keywords: laparoscopic liver resection; cytokine release
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laparoscopic liver resection

SUMMARY:
The purpose of this study is to determine whether the postoperative insulin resistance and cytokine release would be attenuated in laparoscopic compared with open liver resection.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* left hemihepatectomy(liver resection)
* left lateral sectionectomy(liver resection)

Exclusion Criteria:

* Patients with diabetes mellitus
* drug abuse
* BMI >24 or <18

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
postoperative insulin resistance calculated by serum insulin and blood glucose | within the first 72hrs after operation
  At baseline prior to surgery, and 3hr, 12hr, 24hr, 72hrs after operation, blood glucose and insulin was measured.
  Insulin resistance is assessed by the HOMAIR(homeostatic model assessment of insulin resistance) score which is calculated through the mathematic formula: HOMAIR= FI ×FG/22.5, where FI= fasting serum insulin(μU/mL), FG= fasting plasma glucose (mmol/L), and 22.5 is a constant.

SECONDARY OUTCOMES:
cytokine changement including IL-1β, IFN-γ, IL-4 and IL-10 before and after operation | within 5 days after operation
  At baseline before operation and 0, 3hr, 12hr, 24hr, D3, D5 after operation, duplicated samples were drawn to analyze serum IL-1β, IFN-γ, IL-4 and IL-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China